CLINICAL TRIAL: NCT03405584
Title: Efficacy of High Dose of Dual Therapy Plus Bismuth for Helicobacter Pylori Treatment：a Randomized Clinical Trial
Brief Title: High Dose of Dual Therapy Plus Bismuth for Helicobacter Pylori Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rjkls2017196
Record Dates: First submitted 2018-01-13; First posted 2018-01-23 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-01

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Therapy
MeSH Terms: interventions — Esomeprazole; Amoxicillin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bismuth Plus Dual Therapy (Experimental): Esomeprazole 40mg bid, Amoxicillin 1.0g tid and Bismuth Potassium Citrate 600mg bid for 14 days.
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin; Drug: Bismuth Potassium Citrate
- Dual Therapy (Active Comparator): Esomeprazole 40mg bid and Amoxicillin 1.0g tid for 14 days.
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin

INTERVENTIONS:
Drug: Esomeprazole — Proton pump inhibitor
Drug: Amoxicillin — Antibiotic for H. pylori eradication
Drug: Bismuth Potassium Citrate — Gastric mucosal protective drug with anti-H. pylori effect
  Arms: Bismuth Plus Dual Therapy

SUMMARY:
Dual therapy for Helicobacter Pylori including a proton pump inhibitor (PPI) and amoxicillin. Amoxicillin has low resistance rate as well as low percentage of side effects. No trial has examined the the efficacy of high dose of dual therapy plus bismuth for H. pylori treatment.This study is designed to evaluate the efficacy and safety of the addition of bismuth to high dose of dual therapy for H. pylori eradication.

ELIGIBILITY:
Inclusion Criteria:

* Participants with non-ulcer functional dyspepsia or peptic ulcer disease
* Ability and willingness to participate in the study and to sign and give informed consent
* Confirmed H. pylori infection

Exclusion Criteria:

* Less than 18 years old
* With previous gastric surgery
* Major systemic diseases
* Pregnancy or lactation
* Allergy to any of the study drugs Administration of antibiotics, bismuth, antisecretory drugs in 8 weeks prior to inclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).

SECONDARY OUTCOMES:
Rate of adverse effects | Within 7 days after completion of therapy.
  The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or "severe" (causing considerable interference with daily activities).
Compliance rate | Within 7 days after completion of therapy.
  Compliance was defined as poor when they had taken less than 80% of the total medication.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, M.D, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No